CLINICAL TRIAL: NCT03998956
Title: Study of High-density Mapping-guided bOx Isolation and subsTrate Ablation for Persistent Atrial Fibrillation
Brief Title: High-density Mapping-guided bOx Isolation and subsTrate Ablation
Acronym: HOT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: The Third Xiangya Hospital of Central South University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 3rdxiangya@csu
Record Dates: First submitted 2019-06-25; First posted 2019-06-26 (Actual); Last update posted 2019-07-01 (Actual); Status verified 2019-06

CONDITIONS: Atrial Fibrillation; Atrial Remodeling
Keywords: catheter ablation
MeSH Terms: conditions — Atrial Fibrillation; Atrial Remodeling

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Circumferential PV isolation (Active Comparator): Circumferential PV isolation only
  Interventions: Procedure: CPVI
- Circumferential PV and BOX isolation (Experimental): Circumferential PV and BOX isolation
  Interventions: Procedure: CPVI+BOX
- circumferential PV and BOX isolation with substrate ablation (Experimental): Atrial substrate ablation apart from circumferential PV and BOX isolation
  Interventions: Procedure: CPVI+BOX+SUB

INTERVENTIONS:
Procedure: CPVI — Circumferential PV isolation only
  Arms: Circumferential PV isolation
Procedure: CPVI+BOX — Circumferential PV and BOX isolation
  Arms: Circumferential PV and BOX isolation
Procedure: CPVI+BOX+SUB — Atrial substrate ablation apart from circumferential PV and BOX isolation
  Arms: circumferential PV and BOX isolation with substrate ablation

SUMMARY:
This study evaluates the efficacy of high-density mapping guided atrial substrate ablation for persistent atrial fibrillation. 1/5 of the patients with persistent atrial fibrillation undergo pulmonary veins isolation, 2/5 of them pulmonary veins and box isolation while others undergo atrial substrate ablation apart from pulmonary veins and box isolation.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent signed.
* Age of 18 to 75 years old.
* Persistent or longstanding persistent atrial fibrillation (≥7 days), which is confirmed by Holter in recent six months.
* Willing to have catheter ablation for atrial fibrillation.

Exclusion Criteria:

* Accompanied by serious heart diseases including cardiac valvular diseases, congenital heart diseases, hypertrophic obstructive cardiomyopathy, acute myocardium infarction, unstable anginal pectoris and so on.
* Complete atrioventricular block.
* An acute stroke or contradiction of anti-coagulation.
* Hyperthyroidism.
* Having a history of catheter ablation of atrial fibrillation.
* Left atrial appendage thrombosis confirmed by transesophageal echocardiography.
* Pregnancy or lactation.
* Planning for pregnancy in the near future.
* Myopathy or active liver disease, including patients with sustained increase of serum transaminase of unknown reason and the ones with increased serum transaminase over three times the upper limit of normal.
* Patients of severe renal insufficiency with creatinine clearance lower than 30 ml/min.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2019-08-01 (Estimated); Primary Completion 2021-08-31 (Estimated); Study Completion 2021-08-31 (Estimated)

PRIMARY OUTCOMES:
sinus rhythm maintenance rate | 12 months
  Holter is performed 12months after the procedure and heart rhythm is recorded.

SECONDARY OUTCOMES:
left ventricular ejection fraction | 12 months
  LVEF is evaluated by echocardiography 12months after the procedure.
Stroke or embolic events | 12 months
  History of stroke or embolic events is taken at each follow-up during the period of 12 months after procedure, and if necessary, radiographic examinations will be performed.
Atrial fibrosis | 1 day
  Atrial substrate mapping is performed before and after catheter ablation in one day to evaluate the atrial fibrosis.